CLINICAL TRIAL: NCT04713839
Title: Cross-cultural Adaptation, Reliability, and Validity of Turkish Adult Sensory Processing Scale (ASPS)
Brief Title: Adult Sensory Processing Scale (ASPS) Version of Turkish
Acronym: ASPS
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, ZEYNEP BAHADIR AGCE, Assistant Professor, Uskudar University
Other Study IDs: 61351342-193
Record Dates: First submitted 2021-01-09; First posted 2021-01-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Sensory Processing Disorder
Keywords: Adult Sensory Processing Scale; Reliability and Validity; Psychometrics; Self-report; Adult

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: The participants were invited to the study, then each participant was asked to complete the self-report questionnaires.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — We didn't have an intervention program, we used two questionnaires to evaluate participants.

SUMMARY:
Purpose: Sensory processing is crucial to adaptive behavioral responses in occupational therapy. Nevertheless, information on sensory processing in adults is limited. The Adult Sensory Processing Scale (ASPS) measure behavioral responses indicative of sensory processing in different sensory systems. The aim of the study was to examine the cultural adaptation, reliability, and validity of the ASPS Turkish (ASPS-T).

DETAILED DESCRIPTION:
The current study comprises three parts: cross-cultural adaptation, piloting, and examination of psychometric properties of the ASPS-T. The researcher contacted the developers of the original ASPS and received written permission from the authors to translate it into Turkish. This study was conducted by the Helsinki Declaration and Uskudar University. Clinical Research Ethical Board approved the study. After receiving both written and oral information about the project, all the study participants provided a signed consent form.

Phase 1: The cross-cultural adaptation process Translating the Turkish version of ASPS and the cross-cultural adaptation procedure was carried out under the guidance of Beaton et al. Translation from English to Turkish was performed by two therapists whose mother tongue is Turkish, also have fluent in English. Each of the translations was reviewed by three therapists, after the consensus on the final version, it was turned down by two native English-speaking translators. The final version was compared with the original version to reveal any inconsistencies; no discrepancies were observed. During the translation phase, minimal adjust were made to address linguistic.

Phase 2: Piloting process A pre-assessment was made with a pilot study to explore ASPS-Turkish's cultural harmony. The translated questionnaire was completed by 20 participants to identify any items that were not coherent. Four participants stated that they could not understand the meaning of avoid-kaçınmak, so investigators suggested yaşamamak, and this was accepted by participants. Three participants could not respond to the first item on factor 10, because participants had not traveled by boat or rides before, so that, investigators added the phrase "all types of vehicles" was added to the sentence. All the authors meet to compare the ASPS-T with the original version and assess its suitability after the minimal change, concluding that the current correction did not cause any loss of the meaning of the word. After the changes, pilot study participants evaluated the intelligibility of the scale with a 1 to 5 Likert scale, and confirm the clearness unanimously of them. Therefore, the final version of the ASPS-T which has minor changes was the best representation of the original, and each item was found to be suitable for Turkish patients. The pilot study participants were not included in the sample. After cultural equivalence had been achieved, 405 healthy individuals aged 18 and over were asked to complete the ASPS questionnaire.

Phase 3: Analysis of psychometric properties Exploratory and Confirmatory Factor Analysis (EFA and CFA) were used to measure the construct validity of the instrument, and test-retest analysis (interclass correlation coefficient) and Cronbach's alpha were used to evaluate the reliability of the instrument.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18-64 years, able to read and write, and being healthy

Exclusion Criteria:

* Who has a diagnosis of any disorders that preventing from completing the survey such as cancer or cognitive problems.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants consisted of university students, faculty employees, other employees, and their families. Each participant was invited to participate in the study through a face-to-face interview. After receiving both written and oral information about the project, all the participants who volunteered to take part provided a signed consent form. A total of 460 individuals were called to participate in the study and 55 individuals rejected. Fifty-five of the 405 participants were randomly selected to be re-interviewed, and participants completed the questionnaire again for test re-test protocol.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Adolescent/Adult Sensory Profile | 20 minutes
  Adult Sensory Processing Scale is designed to measure different behavioral response patterns (over-responding, under-responding, and sensory seeking) of specific sensory systems (tactile, proprioceptive, vestibular, auditory, and visual) that are indicative of sensory processing challenges. Sensory responsiveness models related to different sensory systems in adults have been defined by over-responsiveness, under-responsiveness and sensory-seeking patterns similar to those in children. A total of 11 factors and 48 items are defined and the number of questions for each factor is different. All items are rated on a 5-point Likert scale with Never = 1, Rarely = 2, Sometimes = 3, Often = 4, and Always = 5.
Adolescent/Adult Sensory Profile | 18 minutes
  The AASP was developed build on Dunn's sensory processing model and is suitable for aged over 11 years. It consists of 60 items and is used to evaluate individuals' sensory processing skills in daily life. Each item is related to responses to sensory input through six diﬀerent sensory factors that refer to everyday activities, including taste/smell, movement, vision, touch, processing, auditory processing, and activity level. The responses of the participants' sensory stimuli are evaluated in four quadrants: low registration, sensory sensitivity, sensory avoiding, and sensory seeking. The responses record on a Likert scale as almost always, often, sometimes, rarely, and almost never, and the scores of the related items are added to supply the score for each quadrant. The tests to settle the validity and reliability of the AASP were completed by Ucgul et al.

CONTACTS AND LOCATIONS:
Overall Officials: ORKUN ARAN, PHD, Study Chair — Hacettepe University; SEDEF ŞAHİN, PHD, Study Chair — Hacettepe University; ZEYNEP BAHADIR AGCE, PHD, Study Director — Uskudar University
Locations (1):
- Uskudar University, Istanbul, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blanche EI, Parham D, Chang M, Mallinson T. Development of an Adult Sensory Processing Scale (ASPS). Am J Occup Ther. 2014 Sep-Oct;68(5):531-8. doi: 10.5014/ajot.2014.012484. PMID 25184465
- See also: PUBMED LINK — https://pubmed.ncbi.nlm.nih.gov/25184465/